CLINICAL TRIAL: NCT00474136
Title: Open-Label, Randomized, Single Center Study to Compare the Pharmacokinetics of IV Diclofenac Sodium (2 Doses) Versus Oral Diclofenac Potassium in Healthy Adult Volunteers Following Single- and Multiple-Dose Administration
Brief Title: Study to Compare the Pharmacokinetics of IV Diclofenac Sodium (2 Doses)Versus Oral Diclofenac Potassium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Amy Cohen, Javelin Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DFC-PK-006
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Intravenous diclofenac sodium (DIC075V) 18.75 mg
- 2 (Experimental)
  Interventions: Drug: Intravenous diclofenac sodium (DIC075V) 37.5 mg
- 3 (Active Comparator)
  Interventions: Drug: Oral diclofenac potassium 50 mg

INTERVENTIONS:
Drug: Intravenous diclofenac sodium (DIC075V) 18.75 mg — DIC075V 18.75 mg
  Arms: 1
Drug: Intravenous diclofenac sodium (DIC075V) 37.5 mg — DIC075V 37.5 mg
  Arms: 2
Drug: Oral diclofenac potassium 50 mg — Oral diclofenac potassium 50 mg
  Other Names: Cataflam
  Arms: 3

SUMMARY:
The purpose of this study is to assess the pharmacokinetic parameters of intravenous diclofenac sodium (DIC075V) 18.75 mg and 37.5 mg following single- and multiple-dose administration, as compared to oral diclofenac potassium (Cataflam® 50 mg), the approved reference product.

DETAILED DESCRIPTION:
This study is an open-label, three-treatment, six sequence, three-period, single center crossover study to evaluate the pharmacokinetics of intravenous diclofenac sodium DIC075V (18.75 mg and 37.5 mg) versus oral diclofenac potassium (Cataflam® 50 mg) in healthy adult volunteers following single- and multiple-dose administration. Each treatment sequence received 1 dose every 6 hours (for a total of 4 doses per treatment sequence) with a 48-hour washout period between treatment sequences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 55 years of age.

Exclusion Criteria:

* Smoked or used tobacco or nicotine products in the past six months or expects to during the study.
* Known allergy or hypersensitivity to diclofenac, aspirin, or other NSAIDs.
* History of previous and/or present peptic ulceration, GI bleeding or any bleeding diathesis, positive for hepatitis B or hepatitis C or for HIV antibodies, or history of asthma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetic parameters of intravenous diclofenac sodium (DIC075V) 18.75 mg and 37.5 mg following single- and multiple-dose administration, as compared to oral diclofenac potassium (Cataflam® 50 mg), the approved reference product. | Several time points over 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Terri Lunsford, MD, Principal Investigator — Parexel
Locations (1):
- PAREXEL International, Baltimore, Maryland, United States